CLINICAL TRIAL: NCT00523224
Title: A Study of Combined Coronary Artery Bypass Grafting (CABG) and Blood-Borne Autologous Angiogenic Cell Precursors Therapy in Patients With Congestive Heart Failure Due to Ischemic Heart Disease
Brief Title: ACPs Combined With CABG in Patients With CHF
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TheraVitae Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV-002; ACPs-CHF
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-05

CONDITIONS: Congestive Heart Failure
Keywords: Stem cells; Coronary Artery Bypass grafting; Congestive Heart Failure; Coronary Artery Disease; Angiogenesis
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): open lable,single arm , intervention is Angiogenic Cell Precusors(ACPs)
  Interventions: Procedure: Angiogenic Cell Precursors(ACPs) or Vescell TM; Biological: Angiogenic Cell Precusors

INTERVENTIONS:
Procedure: Angiogenic Cell Precursors(ACPs) or Vescell TM — at least 1.5 million of ACPs per one time of treatment
Biological: Angiogenic Cell Precusors — Stem cells type Angiogenic Cell Precusors(ACPs) at least 1.5 million ACPs per each treatment

SUMMARY:
Study title: A Study of Combined Coronary Artery Bypass Grafting (CABG) and Blood-Borne Autologous Angiogenic Cell Precursors Therapy in Patients with Congestive Heart Failure due to Ischemic Heart Disease (ACPs-CHF) Principle Investigator: Kit V. Arom ,M.D.,Ph.D. Deputy Director, Chief Cardio-Thoracic Surgeon, Bangkok Heart Hospital Study objective : To determine the safety and efficacy of injection of blood-borne autologous ACPs into the non-graftable area of the heart of patients with congestive heart failure due to ischemic heart disease Its main goal is evaluation of feasibility and safety of the combined technique. The efficacy of the treatment will be tested in the following trial.

Study Design : Phase I , a single center, a non-randomized, open-label trial to test the safety, of intramyocardium transepicardium administration of ex vivo expanded autologous ACPs administered in combination with CABG operation in patients with congestive heart failure due to ischemic heart disease.

The study is a preliminary training study, under the supervision of the experienced Dr. Patel the U.S. principal investigator.

Study population :

Total expected no. of patients : 5 main selection criteria :

1. Patients with or without signs of congestive heart failure due to ischemic heart disease who had maximal medical treatments. Not suitable to percutaneous intervention
2. All patients must have a recent coronary angiogram. Patients must be able to have OPCAB and then have Angiogenic Cell Precursors(ACPs) in non-graftable and/or infraction regions
3. Age 18 to 80 years
4. MRI demonstrating areas of viable and non-viable myocardium Investigational Product : The patients will be blood drawn 250 ml at D-8 for producting autologous ACPs (VescellTM), On D0 ,at least 1.5 million ACPs with viability >75 % supended in 15 ml sterile cell culture medium will be injected 1 cm apart using a 23 gauge angled needle in 30 spots (0.5 ml /point) to the same patients by direct intramuscular approach at LV during CABG.

The study consists of 4 periods: Screening ( D-14 to-9& D-8,Treatment(D0),Acute Safety follow-up (D1-2& D5-discharge),Chronic follow-up (D30 & D90)period ,total follow-up of each case is 3 months.

Evaluation criteria :

Safety : no.& duration of adverse event & serious adverse event Efficacy :NYHA, 6-minute walking test ,% LVEF by Echocardiography & C-MRI, % infracted scar area on C-MRI , Pro-BNP & 3 months of QoL(SF-36)

DETAILED DESCRIPTION:
Five CAD patients who required CABG with or without congestive heart failure will undergo screening and receiving of ACPs 's injection by direct intramuscular during CABG operation. After that,the patients will come to follow up with investigator at 1 and 3 months post surgery in order to evaluate safety and efficacy of stem cells therapy(ACPs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with or without signs of congestive heart failure due to ischemic heart disease who had maximal medical treatments. Not suitable to percutaneous intervention
2. All patients must have a recent coronary angiogram. Patients must be able to have OPCAB and then have Angiogenic Cell Precursors(ACPs) in non-graftable and/or infraction regions
3. Age 18 to 80 years
4. Male or non-pregnant, non-lactating female
5. MRI demonstrating areas of viable and non-viable myocardium
6. Informed consent obtained and consent form signed

Exclusion Criteria:

1. Prior Cardiac Surgery or Heart Transplantation
2. Patient who received blood transfusions during the previous 4 weeks (to exclude the potential of non-autologous ACPs in the harvested blood).
3. Inability to communicate (that may interfere with the clinical evaluation of the patient)
4. Acute Myocardial infarction < 6 days from acute event
5. Significant valvular disease or after valve replacement
6. Left Ventricular Aneurysm
7. Collagen tissue disease
8. History of Prior Radiation Exposure
9. History of alcohol or drug abuse within 3 months of screening
10. Renal failure (creatinine > 2 mg/dl) or Hemodialysis
11. Hepatic failure or History of Liver Cirrhosis
12. Females who are capable of reproduction and will not take acceptable measures to prevent reproduction during the study.
13. Anemia (lower than 11mg/dl.hemoglobin for female and lower than 12 mg/dl for male)
14. Abnormal coagulation tests normal [platelets, PT (INR), PTT]
15. Stroke within the preceding 3 years
16. Malignancy within the preceding 3 years
17. Concurrent chronic or acute infectious disease
18. Severe concurrent medical disease (e.g., septicemia, HIV-1,2/HBV/HCV infections, insulin-dependent diabetes mellitus, systemic lupus erythematosus, multiple sclerosis, amyotrophic lateral sclerosis)
19. Chronic immunomodulating or cytotoxic drugs treatment
20. Patients who have rectal temp. above 38.40C for 2 consecutive days
21. Patient unlikely to be available for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2006-01; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation criteria | 3 months
Safety : no.& duration of adverse event & serious adverse event | 3 months
Efficacy : EF , NYHA | 3 months
change from baseline to 1 & 3 months of NYHA, 6-minute walking test | 3 months
Change from baseline to 3 months of QoL(SF-36) | 3 months

SECONDARY OUTCOMES:
Efficacy:%EF,NYHA | 3 months
change from baseline to 3 months of % LVEF by Echocardiography & C-MRI | 3 months
change from baseline to 3 months of % infracted scar area on C-MRI | 3 months
change from baseline to 3 months of QoL(SF-36) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kitipan Visudharom, Ph.D.,M.D., Principal Investigator — Bangkok Heart Hospital, 2 Soi Soonvijai 7,New Petchburi Rd.,Bangkok 10310 Thailand
Locations (1):
- Theravitae Co., Tel Viv, P.O. B 4049,Ness Ziona, Israel